CLINICAL TRIAL: NCT04958798
Title: Culturally Centering Medications for Opioid Use Disorder With American Indian and Alaska
Brief Title: Culturally Centering Medications for Opioid Use Disorder With American Indian and Alaska Native Communities
Acronym: CTN-0096
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: University of New Mexico (Other)
Responsible Party: Principal Investigator, Aimee Campbell, Research Scientist, New York State Psychiatric Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #8026
Record Dates: First submitted 2021-07-06; First posted 2021-07-12 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Opioid-use Disorder
Keywords: American Indian; Alaska Native; Medications for Opioid-use Disorder; Implementation; Cultural centering
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Culturally Centered MOUD Implementation (Experimental): Culturally centered program-level implementation intervention to increase the use of medications for opioid use disorder in healthcare and treatment settings serving AI/AN communities
  Interventions: Behavioral: Culturally Centered MOUD Implementation Intervention

INTERVENTIONS:
Behavioral: Culturally Centered MOUD Implementation Intervention — Support clinical sites to culturally center the delivery of medications for opioid use disorder through evidence-based implementation strategies tailored to local needs

SUMMARY:
This is a formative research study to test a culturally-centered, program-level implementation intervention to increase the use of medications for opioid use disorder in four healthcare and addiction specialty treatment sites serving American Indian and Alaska Native communities.

DETAILED DESCRIPTION:
This is a formative research study to test a culturally-centered, program-level implementation intervention to increase the use of medications for opioid use disorder (MOUD) in four healthcare and addiction specialty treatment sites serving American Indian and Alaska Native communities. The study design is a cluster randomized stepped wedge implementation trial with two steps, and two sites per step (N=4 sites). Study design and methods are informed by the Consolidated Framework for Implementation Research (CFIR) and the RE-AIM framework (Reach, Effectiveness, Adoption, Implementation, Maintenance). The primary outcome of the trial is the number of consumers with OUD initiated onto MOUD (i.e., buprenorphine, extended-release naltrexone, or methadone) in the 6 months after intervention delivery (compared to the 6 months before intervention delivery) - capturing implementation intervention Reach. The primary outcome will be measured at the end of the six-month implementation stage and compared to the pre-intervention observation phase (prior to delivery of the implementation intervention). Primary data collection will use de-identified data from the electronic medical records (EMR) at each site beginning with data from the six months prior to intervention delivery for Step 1 sites and 12 months prior for Step 2 sites. For Step 1 sites, some secondary outcomes will also be assessed during the sustainment stage (the six months following implementation). As part of the study, consumers with OUD will be asked to participate in additional assessments and provide informed consent. Enrolled consumer participants will be asked to complete four assessment visits (baseline, week 4, week 8, and week 12) to collect comprehensive information about mental health, cultural connectedness and spirituality, social functioning, and experiences with and acceptability of OUD treatment. Providers at each clinical site will also be asked to complete surveys at three time points to assess attitudes, knowledge, and readiness related to MOUD.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* English comprehension and proficiency
* Receiving services at a participating study site
* Meet criteria for a current opioid use disorder
* Self-identify as American Indian or Alaska Native
* Willing to have program data linked to assessment data
* 18 years or older

Exclusion Criteria:

* participation in research assessments contraindicated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Actual)
Dates: Start 2021-12-20 (Actual); Primary Completion 2024-12-13 (Actual); Study Completion 2025-01-16 (Actual)

PRIMARY OUTCOMES:
# consumers with OUD initiated onto MOUD | 6 months
  number of consumers with OUD initiated onto MOUD in the 6 months after intervention delivery compared to pre-intervention

SECONDARY OUTCOMES:
# consumers with OUD offered MOUD | 6 months
  number of consumers with OUD offered MOUD in the 6 months after intervention delivery compared to pre-intervention
# consumers screened for OUD of the overall # of new consumers | 6 months
  number of consumers screened for OUD of the overall number of new consumers in the 6 months after intervention delivery compared to pre-intervention
# consumers with OUD retained in care for at least three months | 6 months
  number of consumers with OUD retained in care for at least three months in the 6 months after intervention delivery compared to pre-intervention

CONTACTS AND LOCATIONS:
Locations (3):
- United States (3):
  - Southcentral Foundation, Anchorage, Alaska
  - Native American Community Clinic, Minneapolis, Minnesota
  - Missouri Breaks, Eagle Butte, South Dakota

IPD SHARING:
Plan to Share IPD: No
Data from this study is owned by participating Tribal clinical sites; any use of IPD requires Tribal (or equivalent organizational) approval.

REFERENCES:
- [Background] Hirchak KA, Nadeau M, Vasquez A, Hernandez-Vallant A, Smith K, Pham C, Oliver KA, Baukol P, Lizzy K, Shaffer R, Herron J, Campbell ANC, Venner KL; CTN-0096 Collaborative Board. Centering culture in the treatment of opioid use disorder with American Indian and Alaska Native Communities: Contributions from a National Collaborative Board. Am J Community Psychol. 2023 Mar;71(1-2):174-183. doi: 10.1002/ajcp.12620. Epub 2022 Aug 23. PMID 35997562
- [Derived] Paschen-Wolff MM, Campbell ANC, Vasquez A, Kessler J, Jansen K, Arnatt CP, Rosa C, Hebden HM, Radin S, Stately A, Shaw J, Kennedy F, Matthews AG, Venner KL. Conducting an implementation intervention study with American Indian and Alaska Native communities: Methodological considerations. Contemp Clin Trials. 2025 Aug;155:107992. doi: 10.1016/j.cct.2025.107992. Epub 2025 Jun 20. PMID 40544955